CLINICAL TRIAL: NCT06782659
Title: A Phase 1 Pharmacokinetic/Bioequivalence Study of 100 Mg of HEZKUE® (ASP-001, Sildenafil) Versus 100 Mg of VIAGRA® (Sildenafil) Film-Coated Tablets Under Fasted Conditions in Healthy Adult Male Subjects
Brief Title: Study to Compare the Effects of Viagra® Vs Hezkue® in Healthy Fasted Male Participants.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aspargo Labs, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ASP-001-005-BE
Record Dates: First submitted 2025-01-08; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction; Viagra; Sildenafil; bioequivalence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm 1 - ASP-001 and Viagra (Experimental): Participants receive 100 mg of ASP-001 followed by a 6 day washout before receiving 100 mg of Viagra
  Interventions: Drug: ASP-001; Drug: Viagra; Device: ASP-001
- Arm 2 - Viagra and ASP-001 (Experimental): Participants receive 100 mg of Viagra followed by a 6 day washout before receiving 100 mg of ASP-001
  Interventions: Drug: ASP-001; Drug: Viagra; Device: ASP-001

INTERVENTIONS:
Drug: ASP-001 — Oral liquid suspension of sildenafil
Drug: Viagra — Sildenafil film-coated tablet
Device: ASP-001 — Bottle/pump containing ASP-001 suspension

SUMMARY:
The objective of this phase 1, open-label, single-center, two-way crossover trial is to evaluate the pharmacokinetics (PK), safety, and tolerability of 100 mg ASP-001 oral liquid suspension versus 100 mg Viagra (sildenafil citrate) tablets in fasted, healthy male volunteers

DETAILED DESCRIPTION:
This is a Phase 1, open-label, single-center, two-way crossover study to evaluate the pharmacokinetics (PK), bioequivalence (BE), safety, and tolerability of ASP-001 (oral liquid suspension of sildenafil) compared to Viagra (sildenafil film-coated tablet) under fasted conditions in 56 healthy adult male participants.

The study aims to demonstrate bioequivalence between the ASP-001 and Viagra formulations and to evaluate whether the absorption rate of ASP-001 is superior to that of Viagra. Additionally, the study assesses the tolerability of ASP-001, including potential for oral irritation, dizziness, or headache.

Participants are randomized to one of these two sequences:

* Sequence 1: ASP-001 in Period I, Viagra in Period II.
* Sequence 2: Viagra in Period I, ASP-001 in Period II

There is a washout period of 6 days between treatment periods.

Enrollment may be increased at any point in this trial to ensure a minimum of 56 evaluable participants.

ELIGIBILITY:
Inclusion Criteria:

* The participant must be informed of the nature of the study and voluntarily agree to participate by signing an informed consent form prior to any study-specific procedures.
* Participants must be healthy male volunteers aged 18 to 55 years (inclusive) at the time of dosing.
* Participants must have a body mass index between 18.0 and 29.9 kg/m² (inclusive) and a body weight of 50 to 100 kg (inclusive).
* Participants must be judged by the Investigator or designee to be in good general health, as documented by medical history, physical examination, clinical laboratory tests, vital signs, and 12-lead electrocardiogram (ECG). Any deviations from normal ranges must be assessed and deemed not clinically significant by the Investigator or designee.
* Participants must have a creatinine clearance (CrCl) value greater than 80 mL/min, as calculated by the Cockcroft-Gault equation.
* Participants must agree to practice an acceptable method of contraception as outlined in the protocol.

Exclusion Criteria:

* Unwillingness or inability to follow the procedures specified by the protocol.
* Participant received any investigational drug/product within 30 days prior to the first dose.
* History of significant renal, hepatic, cardiovascular (including orthostatic hypotension), psychiatric, neoplastic, inflammatory, infectious, diabetes mellitus, or other disease which, in the opinion of the Investigator, represents a safety risk for taking part in the study.
* Presence of any clinically significant results from laboratory tests, vital signs assessments, and electrocardiograms, as judged by the Investigator and/or designee.
* Any degree of hepatic impairment based on liver function testing (abnormal ALT, AST, bilirubin, alkaline phosphatase, prothrombin time and international normalized ratio during screening).
* Demonstrates a reactive screen for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody.
* Reports a clinically significant illness during the 28 days prior to first dose (as determined by the Investigator and/or designee).
* Subjects with known hypersensitivity to sildenafil or any component in the study medication, such as peppermint oil.
* Reports a history of clinically significant allergies including food or drug allergies as judged by the Investigator.
* History of drug abuse within the previous year, or a positive drug screen (amphetamines, barbiturates, benzodiazepines, cannabinoids, Cocaine, Opiates, Phencyclidine, 3,4-methylenedioxymethamphetamine (MDMA)) at screening and/or Day -1.
* Regular alcohol consumption of >15 units per week, with one unit being equivalent to 330mL of beer or 125 mL of wine or 25 mL to 40 mL of ≥ 40% spirits, or a positive alcohol breathalyzer test at screening and/or Day -1.
* Reports use of CYP enzyme inhibitors within 14 days prior to Period 1 dosing.
* Reports use of CYP enzyme inducers or St. John's Wort within 28 days prior to Period 1 dosing.
* Use of prescription or non-prescription drugs, including individual vitamins, herbal and dietary supplements within seven days or five half-lives, whichever is longer, unless in the opinion of the Investigator and Sponsor's medical monitor the medication is not expected to interfere with the study procedures or compromise subject safety (occasional use of acetaminophen, naproxen, and ibuprofen are allowed).
* Blood donation or significant blood loss within 3 months before screening. All volunteers will be advised not to donate blood for 30 days after completing the study.
* Reports donating plasma (e.g., plasmapheresis) within 14 days prior to first dose. All volunteers will be advised not to donate plasma for 30 days after completing the study.
* Demonstrates, in the opinion of study staff, inadequate veins or veins unsuitable for repeated venipuncture (e.g., veins difficult to locate, access, or puncture; veins with a tendency to rupture during or after puncture).
* Reports difficulty fasting or consuming standardized meals.
* Subjects who have difficulty swallowing.
* Regular use of tobacco (>4 cigarettes per day) or nicotine-containing products within four weeks before screening, or urinary cotinine level indicative of active smoking at screening and/or Day -1
* Major surgery within three months or minor surgery within one month before screening as per the Principal Investigator (PI) judgment.

If, in the opinion of the PI, the subject is not suitable for the study.

* Institutionalized volunteers.
* Reports use of any hormone replacement therapy within 6 months prior to first dose.
* Use of any products containing Seville oranges, grapefruit and pomelo within seven days prior to first dose and for the duration of the study.
* Ingestion of any caffeine/xanthine containing products (coffee, tea, soft drinks, chocolate, energy drinks, etc.), foods containing poppy seeds within 48 hours prior to first dose and for the duration of the study.
* Ingestion of any beverages containing more than 5% fruit juice (fruit drinks, fruit punches, fruit cocktails, fruit-ades, or other products containing 5% or less of fruit juice will be allowed) within 48 hours prior to first dose and for the duration of the study.
* Subject administered COVID-19 vaccine within three days prior to each check-in.
* Subjects with retainers, braces, dentures, partial dentures, and/or tongue piercing.
* Subjects using the following within 14 days of first dose:

  * Antihypertensive medications.
  * PDE5 inhibitors
* Subjects with known hypertension or blood pressure and heart rate outside of the following ranges:

  * Systolic blood pressure: 90 - 140 mmHg
  * Diastolic blood pressure: 50 - 90 mmHg
  * Heart rate at screening: 50 - 100 beats per minute

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cisgender
Enrollment: 56 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Cmax | Baseline and at 24 different timepoints during the 24 hour post-dose
  The PK profile of ASP-001 and Viagra in healthy male subjects. Calculation of maximum plasma concentration (Cmax) over the specified timeframe.
Absorption | Baseline and at several timepoints during the 24 hour post-dose
  To determine if the rate and extent of absorption are similar for 100 mg of ASP-001 administered as 8 pumps of the 25 mg/mL oral liquid suspension of sildenafil compared to 100 mg Viagra (sildenafil) administered in the form of a film-coated tablet.
AUCt | Baseline and at 24 different timepoints during the 24 hour post-dose
  The PK profile of ASP-001 and Viagra in healthy male subjects. Calculation of the area under the plasma concentration versus time curve will be calculated using the linear trapezoidal rule from the zero time point to the last quantifiable concentration (AUCt).
AUCi | Baseline and at 24 different timepoints during the 24 hour post-dose
  The PK of ASP-001 and Viagra in healthy male subjects. The area under the plasma concentration versus time curve from zero to infinity (AUCi) will be calculated by adding the last quantifiable concentration (Ct)/ elimination rate contant (Kel) to AUCt.
Tmax | Baseline and at 24 different timepoints during the 24 hour post-dose
  The PK of ASP-001 and Viagra in healthy male subjects. Calculation of the time of the maximum measured plasma concentration (Tmax). If the maximum plasma concentration occurs at more than one time point, the first is chosen as Tmax.
Kel | Baseline and at 24 different timepoints during the 24 hour post-dose
  The PK of ASP-001 and Viagra in healthy male subjects. Calculation of the terminal elimination rate constant obtained from the slope of the line, fitted by linear least squares regression, through the terminal points of the log (base e) of the concentration versus time plot for these timepoints.
tHalf | Baseline and at 24 different timepoints during the 24 hour post-dose
  PK of ASP-001 and Viagra in healthy male subjects. The half-life will be calculated by the equation tHalf = 0.693/ Kel. Apparent elimination half-life.

SECONDARY OUTCOMES:
Number of participants with oral irritation, dizziness, or headache. | Baseline and different timepoints during the 24 hour post-dose
  To determine the potential of ASP-001 to cause oral irritation, dizziness, or headache. Descriptive summaries (mean, standard deviation (SD), median, minimum, and maximum) of actual values and changes from baseline will be provided.
Number of participants with adverse events | Baseline and at several timepoints during the 24 hours post-dose
  The frequency and type of adverse events reported during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Evolution Research Group, Clinical Pharmacology of Miami (CPMI), Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No